CLINICAL TRIAL: NCT01735981
Title: The Effect of Video Game Biofeedback Modulated Exercise (ViBE)on Dynamic Balance and Gait in Individuals With Huntington's Disease
Brief Title: The Effect of Video Game Exercise on Dynamic Balance and Gait in Individuals With Huntington's Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Anne Kloos (Other)
Responsible Party: Sponsor-Investigator, Anne Kloos, Associate Professor Clinical Health and Rehabilitation Sciences, Ohio State University
Organization: Ohio State University (Other)
Allocation: Non-Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2008H0109
Record Dates: First submitted 2012-11-07; First posted 2012-11-28 (Estimated); Results first posted 2021-08-09 (Actual); Last update posted 2021-08-09 (Actual); Status verified 2021-07

CONDITIONS: Huntington's Disease
Keywords: Huntington's Disease; gait; exercise; balance; video game
MeSH Terms: conditions — Huntington Disease; Motor Activity | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: Participants completed one arm of the study and then crossed over into the other arm of the study
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- video game exercise (Experimental): Video game exercise using Dance Dance Revolution
  Interventions: Other: Video game exercise using Dance Dance Revolution; Other: hand-held video game
- control (Other): hand-held video game control
  Interventions: Other: Video game exercise using Dance Dance Revolution; Other: hand-held video game

INTERVENTIONS:
Other: Video game exercise using Dance Dance Revolution — use of the video-game, Dance, Dance Revolution as an exercise to improve gait and balance
  Other Names: exercise; video-game based exercise
Other: hand-held video game — hand-held video games

SUMMARY:
To examine the benefits of using a video-game, Dance, Dance, Revolution, as an exercise modality to improve gait and balance in individuals with Huntington's disease.

DETAILED DESCRIPTION:
The primary purpose of this study was to determine the effectiveness of a therapist-guided Video-game Biofeedback Modulated Exercise (ViBE) program administered via Dance Dance Revolution to improve dynamic balance, gait and mobility in individuals with Huntington's Disease. Secondary aims were to explore whether the ViBE intervention would improve quality of life, fall risk, and neuropsychological functions. The investigators hypothesized that the video-game program would lead to greater improvements in walking, dynamic balance, quality of life, fall risk, and neuropsychological function than a control handheld video game program. Since motivation is essential to the long-term maintenance of an exercise program the investigators were also interested in finding out how successful people with Huntington's Disease were at playing Dance Dance Revolution, what their perceptions were of playing the game, and whether they thought that it was beneficial

ELIGIBILITY:
Inclusion Criteria:

* adults 18 - 79 with a diagnosis of Huntington's disease

Exclusion Criteria:

* cannot walk 10 feet without assistance, any other neurologic condition

Ages: 18 Years to 79 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2008-06; Primary Completion 2010-11 (Actual); Study Completion 2012-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Deb Kegelmeyer, DPT, MS, Principal Investigator — Ohio State University; Anne Kloos, PT, PhD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University Atwell Hall, Columbus, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Dance Dance Revolution Exercise, Then Hand Held Video Game (Control): Participants first completed the video game exercise using Dance Dance Revolution: use of the video-game, Dance, Dance Revolution as an exercise to improve gait and balance. Then participated in a hand held video game as the control activity.
- Hand Held Video Game (Control), Then Dance Dance Revolution Exercise: Individuals first participated in the control group: a hand-held video game. Then completed the video game exercise using Dance Dance Revolution: use of the video-game, Dance, Dance Revolution as an exercise to improve gait and balance.
Period: Allocated
Arm/Group | Dance Dance Revolution Exercise, Then Hand Held Video Game (Control) | Hand Held Video Game (Control), Then Dance Dance Revolution Exercise
Started | 13 | 11
Completed | 11 | 8
Not Completed | 2 | 3
Period: Crossed Over
Arm/Group | Dance Dance Revolution Exercise, Then Hand Held Video Game (Control) | Hand Held Video Game (Control), Then Dance Dance Revolution Exercise
Started | 11 | 7 (N=1 lost to cross over before DDR intervention)
Completed | 11 | 7
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dance Dance Revolution Exercise, Then Hand Held Video Game (Control) | Hand Held Video Game (Control), Then Dance Dance Revolution Exercise | Total
Number analyzed (Participants) | 13 | 11 | 24
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.9 (13) | 50 (16.4) | 51.6 (14.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 6 | 15
  Male | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: forward velocity.
Time Frame: 6 weeks
Population: GAITRite outcome data was eliminated for one participant who consistently exhibited an abnormal gait during testing sessions on the walkway that did not reflect his usual walking pattern. One participant could not walk backward. Thus, 17 participants were included in the GAITRite analysis (n = 16 for backward condition).
Measure: Mean (Standard Deviation); unit: meters per second
Groups:
- Dance Dance Revolution Exercise: All participants who completed the video game exercise using Dance Dance Revolution either in the first 6 weeks of the study or the second 6 weeks.
- Hand Held Video Game (Control): All participants that completed the hand-held video game control group for the first 6 weeks or the second 6 weeks of the study.
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
meters per second | 1.289 (0.47) | 1.292 (0.47)

2. Secondary Outcome: Tinetti Mobility Test
Description: Observation of gait and balance with quantifiable 16-item assessment with an ordinal scale of 0-2 for up to a total score of 32, with higher scores indicating better performance. It is reliable and predicts falls among those with Parkinson's disease and Huntington's disease.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 18 | 18
score on a scale | 22.94 (4.23) | 22.61 (3.29)

3. Secondary Outcome: Four Square Step Test
Description: Examines ability to step over an object in multiple directions and is timed. Participants are instructed to step over a cane into each square in a specific order. Faster times indicate better balance. It has been shown to predict falls in the elderly.
Time Frame: 6 weeks
Population: Loss of one participant in Four-Square Step Test due to incomplete data
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
seconds | 10.19 (3.77) | 10.02 (7.81)

4. Secondary Outcome: Activities-Specific Balance Confidence Scale
Description: Individuals rate their balance confidence from 1-100 on 16 tasks and total score is the mean; higher scores indicate greater confidence and lower fall risk. The Activities-Specific Balance Confidence Scale is reliable and valid in elderly and neurological populations.
Time Frame: 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 18 | 18
score on a scale | 78.40 (15.64) | 77.56 (15.24)

5. Secondary Outcome: World Health Organization Quality of Life
Description: This questionnaire is a measure of quality of life addressing 4 domains including physical, psychological, social, and environment health. Responses on 26 items are on a five-point scale (from 1 = very dissatisfied to 5 = very satisfied) and each item is added to achieve a total score for each domain. The mean score for each domain is calculated then multiplied by 4 to get the domain score which are then transformed to a scaled score of 0-100 comparable to the original WHOQOL-100 therefore a total score between 0-400 with high scores indicating better quality of life. The WHOQOLBref has good reliability and validity.
Time Frame: post intervention and post hand-held game, each lasts 6 weeks
Population: Loss of one participant for the WHOQOL-Bref due to incomplete data
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Video Game Exercise | Control
Number analyzed (Participants) | 17 | 17
score on a scale | 286 (67.96) | 294 (58.96)

6. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: forward stride length.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
cm | 123.35 (35.23) | 123.11 (35.9)

7. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: forward swing percent.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of gait cycle spent in swing
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
percentage of gait cycle spent in swing | 36.82 (3.64) | 36.01 (4.33)

8. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: forward double support percent.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of gait cycle in double support
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
percent of gait cycle in double support | 25.83 (7.36) | 28.34 (8)

9. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: forward heel to heel base of support.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
cm | 12.37 (5.14) | 12.69 (5.41)

10. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: backwards velocity.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 16 | 16
meters per second | 0.81 (0.41) | 0.83 (0.42)

11. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: backwards stride length.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 16 | 16
cm | 81.09 (31.78) | 83.44 (32.6)

12. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: backwards swing percent.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of gait cycle spent in swing
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 16 | 16
percentage of gait cycle spent in swing | 37.24 (4.05) | 35.83 (4.37)

13. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: backwards double support percent.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percent of gait cycle in double support
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 16 | 16
percent of gait cycle in double support | 26.43 (10.54) | 30.71 (9.44)

14. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: backwards heel to heel base of support.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 16 | 16
cm | 20.61 (5.71) | 21.28 (5.41)

15. Primary Outcome: Gait Parameters
Description: utilized GAITRite to obtain spatiotemporal measures of gait: obstacle velocity.
Time Frame: 6 weeks
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: meters per second
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
Number analyzed (Participants) | 17 | 17
meters per second | 1.16 (0.49) | 1.14 (0.43)

ADVERSE EVENTS:
Time Frame: Course of the time from when the participant was enrolled in the study (8-12 weeks)
Groups:
- Dance Dance Revolution Exercise: All participants who were initially enrolled into the group with the video game exercise using Dance Dance Revolution either in the first 6 weeks of the study or the second 6 weeks.
- Hand Held Video Game (Control): All participants that who were initially enrolled into the control group with the hand-held video game control for the first 6 weeks or the second 6 weeks of the study.
Arm/Group | Dance Dance Revolution Exercise | Hand Held Video Game (Control)
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/18
Other Adverse Events (participants affected / at risk) | 0/24 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No